CLINICAL TRIAL: NCT05758415
Title: A Randomized, Parallel-group, 24 Week, Double-blind, Placebo-controlled, Multicenter Phase 3 Study to Assess the Efficacy and Safety of Secukinumab Compared to Placebo in Adult Patients With Active Rotator Cuff Tendinopathy
Brief Title: Study of Efficacy and Safety of Secukinumab in Participants With Moderate-severe Rotator Cuff Tendinopathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Project discontinued to prioritize other key programs in portfolio
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457O12302; 2022-502080-38-00 (Other: EU CT Number)
Record Dates: First submitted 2023-02-01; First posted 2023-03-07 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Moderate to Severe Rotator Cuff Tendinopathy; Adult; Unilateral; Refractory to standard of care
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, site personnel, persons performing the assessments and participants remained blinded through the Week 24 final database lock. The Novartis clinical trial and submission teams remained blinded to the identity of the treatment from the time of randomization until the Week 16 database lock (for the primary endpoint analysis). The following methods were utilized for blinding: (1) Randomization data were kept strictly confidential until the time of unblinding and were not accessible by anyone else involved in the study with the following exceptions: bioanalyst; (2) the identity of the treatments was concealed by the use of study treatments that were all identical in packaging, labeling, schedule of administration, and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Participants received secukinumab 300 mg at randomization (baseline visit) and Weeks 1, 2, 3, 4, 8, and 12.
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Participants received placebo at randomization (baseline visit) and Weeks 1, 2, 3, 4, 8, and 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — 2 X secukinumab 150 mg / 1 mL as solution for subcutaneous (s.c.) injection
  Other Names: AIN457
  Arms: Secukinumab
Drug: Placebo — 2 X placebo / 1 mL as solution for s.c. injection
  Arms: Placebo

SUMMARY:
The purpose of the present study was to assess the efficacy of secukinumab 300 mg s.c. (subcutaneous) compared to placebo, each in combination with standard of care, in improving signs, symptoms and physical function in participants with moderate to severe rotator cuff tendinopathy (RCT), using a randomized, double-blind, placebo controlled, parallel group design to minimize bias.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled Phase III study, stratified by tear status (no tear/ partial tear) in participants with moderate to severe rotator cuff tendinopathy (RCT), experiencing active disease from at least 6 weeks to 6 months at baseline, and were refractory to standard of care (non-steroidal anti-inflammatory drug [NSAIDs] and course of physiotherapy) over a period of 8 weeks.

The study was terminated due to the project being discontinued in order to prioritize other key programs in the portfolio. Due to the early termination and small sample size, the analysis by tear status stratification was not performed.

The study duration was up to 32 weeks, consisting of a screening period lasting up to 8 weeks (inclusive of a mandatory 2-week run-in period), a 16-week treatment period with last dose administered at Week 12, and an 8-week safety follow-up period. The primary endpoint assessment was at Week 16, and the safety follow-up data collection was through to Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral rotator cuff tendinopathy with ≥ 6 weeks to ≤ 6 months symptom duration at baseline.
2. Nocturnal pain in shoulder on at least 3 out of 7 nights in the week prior to baseline or "positive painful arc test" on examination.
3. Total WORC percentage score ≤ 40 at the screening and baseline visits.
4. Average weekly (i.e., the average of the 7 scores taken once a day) numerical rating scale (NRS) pain score of ≥5 during the past 7 days prior to the baseline visit.
5. Refractory to standard of care: non-steroidal anti-inflammatory drug (NSAIDs) course as per local standard practice (if not intolerant or contraindicated) and a course of physiotherapy over a period of 8 weeks.
6. Participant agreed to remain on stable NSAID dosage regimen (if not intolerant or having contraindications; NSAID dose was permitted to be reduced, but not increased above dose established at run-in) and physiotherapy regimen from run-in period until End of Study (EOS).
7. Presence of tendinopathy in the affected shoulder on a centrally read MRI (Magnetic Resonance Imaging), with the following conditions: with no tear or partial tear (maximum 50% tendon thickness; anteroposterior (AP) length maximum 10 mm)

Exclusion Criteria:

1. Rheumatological and non-rheumatological inflammatory diseases, including but not limited to polymyalgia rheumatica (PMR), psoriatic arthritis (PsA), axial spondyloarthritis (AS: ankylosing spondylitis, nr-axSpA: non-radiographic axial spondyloarthritis), psoriasis (PsO), and rheumatoid arthritis (RA); fibromyalgia or severe pain disorder unrelated to the target shoulder; gout; and systemic lupus erythematosus.
2. Rheumatoid factor (RF) or anti-cyclic citrullinated peptide (anti-CCP) antibodies positive at screening.
3. Oral, intramuscular or intravenous (i.v.) corticosteroid treatment within the last 12 weeks prior to randomization, or presence of any condition that might require intermittent corticosteroid use.
4. Lack of compliance with adhering to NSAID (unless intolerant or contraindicated) and physiotherapy regimen during run-in period.
5. Positive painful arc test result in contralateral shoulder
6. Inability or unwillingness to undergo MRI of the shoulder (e.g., participants with pacemakers, or metal fragments/foreign objects in the body that were not compatible with performing an MRI) to fulfill eligibility criteria (unless centrally read MRI images acquired within 3 months of baseline could be provided and the quality of images was deemed sufficient).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (4):
  - Horizon Clinical Research, La Mesa, California
  - Medvin Clinical Research, Van Nuys, California
  - Conquest Research, Winter Park, Florida
  - LV Research, Las Vegas, Nevada
- China (6):
  - Novartis Investigative Site, Wuhan, CHN
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Shanghai
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Siena, SI
- Poland (4):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Swidnica
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
- Spain (5):
  - Novartis Investigative Site, Santiago, A Coruna
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 272 participants were screened in this study, of which 212 discontinued prior to randomization.
Period: Overall Study
Arm/Group | Secukinumab | Placebo
Started | 30 | 30
Completed | 28 | 24
Not Completed | 2 | 6
Not completed — Subject Decision | 2 | 5
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomized set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (9.74) | 49.5 (9.62) | 48.5 (9.65)
Age, Customized [Number; unit: participants]
  25 - < 45 years | 13 | 9 | 22
  45 - <= 65 years | 17 | 21 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 19 | 24 | 43
  Black or African American | 1 | 0 | 1
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Western Ontario Rotator Cuff Index (WORC) Physical Symptom Domain (PSD) Score at Week 16
Description: The WORC PSD is a sub-domain of the WORC Patient-Reported Outcome (PRO) and comprises 6 questions that capture the key symptoms experienced by participants with rotator cuff tendinopathy (RCT) relating to pain, weakness, stiffness, and mechanical symptoms. The raw score was converted to a scale of 0 to 100, where 0 represents the most symptomatic score, and 100 represents no symptoms.
Time Frame: At Week 16
Population: The full analysis set included all participants from the randomized set to whom study treatment was assigned. Number analyzed is the number of participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale | 30.90 (19.250) | 28.69 (27.320)

2. Secondary Outcome: Change From Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) - Short Form (SF) Upper Extremity Score
Description: PROMIS-SF Upper Extremity measures self-reported capability of physical function. Participants were asked a series of 7 questions rating their ability to perform a range of physical activities related to daily life that would be impacted by shoulder function. Each response was scored from 1 (unable to do) to 5 (without any difficulty). The responses for the 7 questions were added to the total raw score ranging from 7 (worst) to 35 (best) and converted to a T-score with a range from 16.3 (worst outcome) to 58.2 (best outcome), which was used for the analysis. Therefore, the theoretical range for the value for change from baseline for converted T-scores was between -41.9 to 41.9. A positive change from baseline indicated a better outcome.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 28 | 23
score on a scale | 7.56 (6.776) | 8.48 (9.744)

3. Secondary Outcome: Percentage of Participants Who Achieved an Improvement (Increase) of at Least 40 Points From Baseline in the WORC PSD Score at Week 16
Description: as for outcome 1
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants | 28.6 | 36.4

4. Secondary Outcome: Percentage of Participants Who Achieved an Improvement (Increase) of at Least 50 Points From Baseline in the WORC Total Score
Description: The WORC is a patient-reported outcome tool, uniquely developed for rotator cuff conditions. The WORC is self-administered and consists of 21 items divided into five domains: physical symptoms, sport/recreation, work function, lifestyle function, and emotional function. The raw score was converted to a scale of 0 to 100, where 0 represents the most symptomatic score, and 100 represents no symptoms.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 28 | 24
percentage of participants | 28.6 | 29.2

5. Secondary Outcome: Percentage of Participants Who Achieved an Improvement (Increase) of at Least 40 Points From Baseline in the WORC PSD Score at Week 24
Description: as for outcome 1
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 21 | 21
percentage of participants | 42.9 | 33.3

6. Secondary Outcome: Change From Baseline in WORC PSD Score at Week 24
Description: as for outcome 1
Time Frame: At Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 21 | 21
score on a scale | 35.79 (21.374) | 27.36 (27.663)

7. Secondary Outcome: Secukinumab Serum Concentrations
Description: Pharmacokinetic parameters (measures of treatment exposure) were evaluated in all participants, with moderate to severe RCT, treated with secukinumab 300 mg s.c.
Time Frame: Day 1 and Weeks 4 and 16
Population: The safety set included all participants who took at least one dose of study treatment during the treatment period. Number analyzed is the number of participants with available data at that timepoint.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Secukinumab
Number analyzed (Participants) | 29
μg/mL
  Day 1 | 0.00 (0.00)
  Week 4: number analyzed (Participants) | 25
  Week 4 | 90.5 (34.5)
  Week 16: number analyzed (Participants) | 25
  Week 16 | 41.8 (18.1)

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs), by Maximum Severity
Description: Severity: Mild - usually transient in nature and generally not interfering with normal activities; Moderate - sufficiently discomforting to interfere with normal activities; Severe - prevents normal activities.
Time Frame: Up to Week 24
Population: The safety set included all participants who took at least one dose of study treatment during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 30 | 30
percentage of participants
  Mild | 20.0 | 26.7
  Moderate | 10.0 | 10.0
  Severe | 0 | 3.3

9. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Laboratory Parameters
Description: Laboratory parameters included alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, albumin, amylase, calcium, creatinine, bilirubin, glucose, lactate dehydrogenase, lipase, magnesium, phosphate, potassium, sodium, urate, and urea nitrogen.
Time Frame: Up to Week 24
Population: The safety set included all participants who took at least one dose of study treatment during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 30 | 30
percentage of participants | 0 | 0

10. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included sitting systolic blood pressure, sitting diastolic blood pressure, and sitting pulse rate.
Time Frame: Up to Week 24
Population: The safety set included all participants who took at least one dose of study treatment during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 30 | 30
percentage of participants | 0 | 0

11. Secondary Outcome: Percentage of Participants With Binding and Neutralizing Anti-drug Antibodies
Time Frame: At Day 1 and Week 16
Population: The safety set included all participants who took at least one dose of study treatment during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 30 | 30
percentage of participants
  Day 1 | 0 | 0
  Week 16 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported up to a maximum duration of 24 weeks.
Arm/Group | Secukinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=30) | Placebo (N=30)
COVID-19 (Infections and infestations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT05758415/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT05758415/SAP_001.pdf